CLINICAL TRIAL: NCT00056264
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled Parallel Group, Dose Finding Study Evaluating the Safety and Efficacy of Infliximab Administration in Symptomatic Subjects With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Study of Safety and Efficacy of Infliximab (Remicade) in Patients With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004795
Record Dates: First submitted 2003-03-07; First posted 2003-03-10 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-04

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD
Keywords: Chronic obstructive pulmonary disease; COPD; Infliximab; Remicade
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Infliximab

INTERVENTIONS:
Drug: Infliximab

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of infliximab (Remicade) in patients with Chronic Obstructive Pulmonary Disease (COPD). Infliximab (Remicade) targets specific proteins in the body's immune system to help control the development of inflammation to help reduce painful disease.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a smoking-related inflammatory lung disease that results in reduced lung function, causing the symptoms or problems that you have when breathing. COPD includes both chronic bronchitis and emphysema. The symptoms of COPD are cough, sputum (phlegm) production, breathlessness, and wheezing. Advanced disease may also involve changes in appetite and weight loss. The drug used in this study is called Remicadeâ, and the active component is called infliximab. Infliximab binds to and blocks the activity of a naturally occurring substance in the body called tumor necrosis factor alpha or TNFa, which may be associated with inflammation and a decrease in lung function.The purpose of this study is to evaluate the safety and effectiveness of infliximab in the treatment of patients with symptoms of moderate to severe COPD.Patients will be receive infusions of either placebo, 3 mg/kg infliximab or 5mg/kg infliximab at weeks 0, 2, 6, 12, 18, and 24.Safety evaluations will be performed at specified intervals throughout the study and will consist of laboratory tests, vital signs (such as blood pressure), physical examinations and the occurrence and severity of adverse events as well as other study specific procedures. Patients will receive infusions of either placebo, 3 mg/kg infliximab or 5mg/kg infliximab at weeks 0, 2, 6, 12, 18, and 24.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have moderate or severe COPD
* Patients must have at least one episode of COPD-related symptoms (eg, cough, sputum production, shortness of breath) within 2 months prior to screening Exclusion Criteria:
* Patients must not have asthma as main component of obstructive airway disease
* Patients must not have had a moderate or severe exacerbation of COPD within previous 1 month

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2002-12; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Chronic Respiratory Questionnaire (CRQ) total score at week 24

SECONDARY OUTCOMES:
Change in pre-bronchodilator predicted forced expiratory volume in 1 second (FEV1) at week 24 , in 6-minute walk distance at week 24, in health survey (SF-36) physical component summary score at week 24, in Transition Dyspnea Index (TDI) score at week 24

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Result] Rennard SI, Fogarty C, Kelsen S, Long W, Ramsdell J, Allison J, Mahler D, Saadeh C, Siler T, Snell P, Korenblat P, Smith W, Kaye M, Mandel M, Andrews C, Prabhu R, Donohue JF, Watt R, Lo KH, Schlenker-Herceg R, Barnathan ES, Murray J; COPD Investigators. The safety and efficacy of infliximab in moderate to severe chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2007 May 1;175(9):926-34. doi: 10.1164/rccm.200607-995OC. Epub 2007 Feb 8. PMID 17290043
- [Derived] Rennard SI, Flavin SK, Agarwal PK, Lo KH, Barnathan ES. Long-term safety study of infliximab in moderate-to-severe chronic obstructive pulmonary disease. Respir Med. 2013 Mar;107(3):424-32. doi: 10.1016/j.rmed.2012.11.008. Epub 2012 Dec 14. PMID 23246078
- [Derived] Loza MJ, Watt R, Baribaud F, Barnathan ES, Rennard SI. Systemic inflammatory profile and response to anti-tumor necrosis factor therapy in chronic obstructive pulmonary disease. Respir Res. 2012 Feb 2;13(1):12. doi: 10.1186/1465-9921-13-12. PMID 22300528
- See also: A Study of Safety and Efficacy of Infliximab (Remicade) in Patients With COPD — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=155&filename=CR004795_CSR.pdf